CLINICAL TRIAL: NCT06932835
Title: Comparison of Postoperative Analgesic Efficacy of Transversus Abdominis Plane Block (TAP) and Modified Thoracoabdominal Nerve Block (M-TAPA) in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Comparison of Postoperative Analgesic Efficacy of Transversus Abdominis Plane Block (TAP) and Modified Thoracoabdominal Nerve Block (M-TAPA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Muruvvet Taskir Turan, Principal investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-043
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Laparoskopic Cholecystectomy; Transversus Abdominis Plane (TAP) Block; Modified Thoracoabdominal Nerve Block (M-TAPA)
Keywords: remifantanile conception; acute pain; Postoperatif pain
MeSH Terms: conditions — Bites and Stings; Acute Pain | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus Abdominis Plane (TAP) Block (Active Comparator): The patient is placed in the supine position,the injection site is disinfected.The Transversus Abdominis Plane block is performed under ultrasound guidance using a high-frequency linear probe(6-13 MHz)placed sagittally at the midpoint between the costal margin and the iliac crest.On ultrasound, the skin, subcutaneous fat tissue, external oblique muscle, internal oblique muscle, and transversus abdominis muscle are visualized. A 2G, 80 mm block needle is inserted in the same plane as the ultrasound probe.As the needle passes through the muscle layers and fascial planes, a fascial "click" sensation is felt, and the needle tip is advanced under ultrasound guidance in a controlled manner.After the second "click" sensation(the passage through the internal oblique muscle fascia) a test dose of 1 mL is administered to confirm needle tip localization.Once the location is verified, 20 mL of 0.25% bupivacaine is injected into the neurofascial plane. then repeated on the contralateral side.
  Interventions: Drug: Transversus Abdominis Plane (TAP) Block
- Modified Thoracoabdominal Nerve Block (M-TAPA) (Active Comparator): The patient is placed in the supine position, and the injection site is disinfected.Modified Thoracoabdominal Nerve Block To identify the transversus abdominis, internal oblique and external oblique muscles a high-frequency linear ultrasound probe (6-13 MHz) is placed sagittally at the 10th costal margin under USG guidance.After positioning the probe sagittally at the 10th costal margin in the midline, it is angled deeply toward the costochondral angle to visualize the lower costal cartilage.Using an in-plane technique, a 22G, 80 mm block needle is inserted in a cranial direction between the transversus abdominis muscle and the lower surface of the costal cartilage. The needle tip is advanced toward the posterior surface of the 10th costal cartilage, and 20 mL of 0.25% bupivacaine is injected beneath the chondrium while ensuring that the needle tip does not pass beyond the cranial border of the 10th costal cartilage. The same procedure is then repeated on the contralateral side.
  Interventions: Drug: Modified Thoracoabdominal Nerve Block (M-TAPA)

INTERVENTIONS:
Drug: Transversus Abdominis Plane (TAP) Block — Transversus Abdominis Plane (TAP) Block is performed under ultrasound guidance before the surgical procedure and anesthesia induction, with the patient in the supine position.
  Arms: Transversus Abdominis Plane (TAP) Block
Drug: Modified Thoracoabdominal Nerve Block (M-TAPA) — Modified Thoracoabdominal Nerve Block (M-TAPA) is performed under ultrasound guidance before the surgical procedure and anesthesia induction, with the patient in the supine position.
  Arms: Modified Thoracoabdominal Nerve Block (M-TAPA)

SUMMARY:
Laparoscopic cholecystectomy is a frequently performed surgical procedure and is considered the gold standard for treating symptomatic gallstone disease. Although laparoscopic cholecystectomy is considered minimally invasive, it can cause moderate to severe pain in the postoperative period. Poorly controlled early postoperative pain can impair recovery quality and increase the risk of postoperative pulmonary complications as a risk factor for chronic pain development. Multimodal analgesia, including opioids, is used to limit pain following laparoscopic cholecystectomy. However, opioid treatment may lead to side effects such as postoperative nausea and vomiting (PONV), respiratory depression, and constipation.

Nerve blocks provide better pain control, reduce opioid consumption in the postoperative period, and offer advantages such as fewer side effects and a lower risk of pulmonary and cardiac complications.

In our clinic, a multimodal analgesia approach is preferred for patients undergoing laparoscopic cholecystectomy. In addition to intravenous analgesic agents, peripheral nerve blocks are administered based on patient preference (for all eligible and consenting patients).

This study aims to compare the postoperative analgesic efficacy of the Transversus Abdominis Plane (TAP) Block and the Modified Thoracoabdominal Nerve Block with a Pericostal Approach (M-TAPA) in patients undergoing laparoscopic cholecystectomy. Standard analgesic methods are applied to patients who do not consent to peripheral nerve block administration.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* American Society of Anesthesiologists (ASA) physical status I-II-III
* Body mass index 18 to 30 kg/m2
* Elective laparoscopic cholecystectomy surgery

Exclusion Criteria:

* Under 18 and over 65
* ASA score IV and above
* Advanced co-morbidity
* History of bleeding diathesis
* Patient refusing the procedure
* Chronic opioid or analgesic use
* Patients who will operate under emergency conditions
* Block injection site infection
* Known allergy to local anesthetics
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-04-11 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
Pain scores | First 24 hours after surgery
  Pain will be assessed at rest and while movement using the from 0 (no pain) to 10 (worst

SECONDARY OUTCOMES:
Intraoperative remifentanil consumption | During The intraoperatif period
  The amount of remifentanil that patients need to maintain anesthesia during the intraoperative period will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)